CLINICAL TRIAL: NCT05668130
Title: Comparison of Sacrospinous Ligament Fixation and Uterosacral Ligament Suspension for Apical Prolapse Surgery: A Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Tulasa Basnet, Assistant professor, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 394/079/080-IRC
Record Dates: First submitted 2022-12-09; First posted 2022-12-29 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pelvic organ prolapse; Sacrospinous ligament fixation; Uterosacral ligament suspension
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacrospinous Ligament Fixation Arm (Experimental): Women randomized to this arm will undergo sacrospinous ligament fixation for apical suspension procedure during pelvic organ prolapse surgery.
  Interventions: Procedure: Sacrospinous ligament fixation
- Uterosacral Liganemt Suspension Arm (Experimental): Women randomized to this arm will undergo uterosacral ligament suspension for apical suspension procedure during pelvic organ prolapse surgery.
  Interventions: Procedure: Uterosacral Ligament Suspension

INTERVENTIONS:
Procedure: Sacrospinous ligament fixation — Women with stage II or higher pelvic organ prolapse with apical compartment involvement planned for surgical management will be randomised to either sacrospinous ligament fixation arm or uterosacral ligament suspension arm. those raandomized to sacrospinous ligament fixation arm will undergo unilateral (right) sided sacrospinous ligament fixation of apex as a part of pelvic organ prolapse surgery.
  Other Names: SSLF
  Arms: Sacrospinous Ligament Fixation Arm
Procedure: Uterosacral Ligament Suspension — Similarly women randomised to uterosacral ligament suspension arm will undergo modified high uterosacral ligament suspension of apex. Both arms will be followed up in 6 months and 12 months for anatomical and functional outcome.
  Other Names: USLS
  Arms: Uterosacral Liganemt Suspension Arm

SUMMARY:
the main aim of this study is to study the anatomical and functional outcomes of two vaginal apical fixation procedures; sacrospinous ligament fixation and uterosacral ligament suspension, for pelvic organ prolapse surgery.

The participants will be randomized to either of the surgical procedure and will be followed up for one year to study the outcome.

DETAILED DESCRIPTION:
1. Objectives General objective To compare the surgical outcome between SSLF and modified USLS for apical fixation in women undergoing vaginal prolapse surgery Specific objectives 1) To compare the success rate of SSLF and modified USLS for apical fixation at 6 month and one year after vaginal prolapse surgery 2) To evaluate perioperative complications of the two procedures 3) To study the change in pelvic floor disorders symptoms in postoperative period ( 6 months and 12 months) among two groups.
2. Methods 2.1. Recruitment: Women with stage II or higher POP with involvement of apical compartment planned for surgical management will be included in the study. Detailed history will be taken regarding demographic profile like age, parity, menopausal status, mode of previous deliveries, history of smoking, heavy weight lifting. The presenting complaints as well as other associated complaints will be noted. History of previous abdominal or pelvic surgeries will be obtained. For recording the history regarding pelvic floor disorders, PFDI 20 (translated in Nepali language and pretested) will be used. General and systemic physical examination will be performed. The BMI will be noted. The prolapse will be examined and staged according to POP-Q staging system. Cough stress test and ESST will be performed to rule out SUI. The tests will be performed after reducing the prolapse to rule out occult SUI. The intended prolapse surgery as well as necessary concomitant surgeries will be decided by the surgeon. Informed written consent will be obtained from the participants for including into the trial.

2.2. Randomization: The participants will be randomized on 1:1 basis to one of the methods of vaginal apical suspension either SSLF or USLS. Computer generated randomization table will be generated and used for randomization. The patients will be randomized by one of the residents posted in unit who is not involved in the research one day prior to surgery after pre-operative examination and decision for surgery is made.

2.3 Surgical procedures The surgeries will be performed by a team of surgeons with technical competency in both the techniques.

Method of Sacrospinous Ligament Fixation (SSLF):

Women who are randomized to this group will undergo unilateral sacrospinous ligament fixation. For all the women with uterine descent requiring the hysterectomy, vaginal hysterectomy will be performed using standard method. In women with vault prolapse, the apex of the vagina is grasped with Allis forceps. A horizontal incision is given in the apex over previous scar of vaginal vault. The enterocele sac will be dissected off the vaginal mucosa. The sacrospinous ligament will be accessed via posterior approach. A vertical incision will be given in the posterior vaginal wall leaving ~2-3 cm bridge of vaginal mucosa between the incision and the vault. The right pararectal space will be entered by blunt dissection till the sacrospinous ligament is reached. The rectum will be mobilized medially. Once the ischial spine is identified, SSL is palpated by dorsal and medial movement of the fingers. Any fibroareolar tissue present over the ligament will be removed with the swab held in sponge holding forceps. Per rectal examination is performed to rule out rectal injury. For proper visualization of SSL, Breisky-Navratil retractor will be used. A permanent suture Polyster no 1 will be passed through the SSL around 1.5 to 2 cm medial to the ischial spine under direct vision with the help of long needle holder. The other end of the suture is brought out to the right end of vaginal vault and it will be tagged. Another suture will be placed in SSL medial to the previous one and again brought out to the vault towards left end and will be tagged. Anterior repair if needed will be performed. The upper portion of posterior vaginal wall mucosa will be closed. The suspension sutures are then tied so that the vagina comes in contact with the SSL without the bridge of suture in between. Posterior colpoperinorrhaphy will then be performed. If anti-incontinence procedures are needed, will also be performed.

Method of Uterosacral Ligament Suspension (USLS) For all the women with uterine descent requiring the hysterectomy, vaginal hysterectomy will be performed using standard method. The pedicles of the uterosacral ligaments will be tagged. For women with vault prolapse, a horizontal incision will be given at the level of vault. It will be opened and the enterocele sac will be dissected off the vaginal mucosa. The enterocele sac will opened for the intraperitoneal access of uterosacral ligament. The posterior-cul-de-sac will be packed with moist gauze. The remnants of the uterosacral ligaments will be identified medial to the ischial spine. A non-absorbable suture; Polyster no 1 will be passed through the uterosacral ligament at the level of ischial spine. Another suture with the same suture material will be passed through the ligament around 1 cm below the ischial spine. The one end of the suture is passed through the anterior vaginal wall and the other end through the posterior vaginal wall. Same procedure will be repeated on the other side. Anterior colporrhaphy if needed will be performed. The suspension sutures will then be tied. Posterior colpoperineorrhaphy, anti-incontinence procedure if needed will be performed thereafter.

In case the allocated procedure cannot be performed for vault suspension, alternative surgery will be performed. If both the procedures cannot be performed, the procedure for apical suspension will be decided by the operating surgeon. During the surgery, duration of the surgery, intraoperative blood loss, occurrence of urinary or bowel injury will be noted. Cystoscopy will be performed after each surgery to rule out urinary tract injury.

2.4. Follow up After the surgery the patients will be managed in postoperative wards as per the hospital protocol. The duration of catheterization, post-operative hospital stay will be recorded. All women will be taught and advised to perform pelvic floor muscle training (PFMT) at the time of discharge. The postmenopausal women will be prescribed with local estrogen cream. Following the discharge women will be scheduled for follow up in 6 months and one year of surgery. However, if patient experiences any complications, she is advised to follow up immediately. The complication developed will be managed as needed and the event will be recorded. During each follow up, women will be enquired about the symptoms according to PFDI-20, POP-Q examination will be performed.

3. Measurement 3.1. Primary outcome Success rate of SSLF and USLS for apical suspension Success will be defined as absence of any of the following

1. Stage II or greater apical compartment prolapse
2. Awareness of bulge symptoms confirmed by affirmative response to question number 3 of PFDI-20.
3. Need of additional treatment for prolapse (ring pessary, repeat surgery)

4.2. Secondary outcome Perioperative outcomes Duration of surgery Intraoperative blood loss Duration of catheterization Duration of Hospital stay

1. Complications Bladder, ureteric or bowel injury, neurological injury, vascular injury Urinary retention, Vault hematoma, Dyspareunia
2. Change in PFDI-20 score The intraoperative blood loss will be calculated by the change in perioperative hematocrit concentration ( difference between pre-operative hematocrit and hematocrit sent on first postoperative day) using the formula(25); Vloss total = BV X (Hctpreop - Hctpostop) The blood volume will be calculated using the formula(26), BV= k1 x H3 + k2 x W + k3 For females, k1 = 0.3561, k2= 03308 and k3 = 0.1833

5. Adverse events

Adverse event (AE) will be recorded as per Clavein Dindo classification of surgical complications which is as follows:

Grades Definition Grade I Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions. Acceptable therapeutic regimens: drugs like antiemetics, antipyretics, analgesics, diuretics and electrolytes and physiotherapy.

Also includes wound infections opened at the bedside. Grade II Requiring pharmacological treatment with drugs other than such allowed for grade I complications.

Blood transfusions and total parenteral nutrition are also included. Grade III Requiring surgical, endoscopic or radiological intervention Grade III-a: intervention not under general anesthesia Grade III-b: intervention under general anesthesia Grade IV Life-threatening complication (including CNS complications) requiring IC/ICU-management Grade IV-a: Single organ dysfunction (including dialysis) Grade IV-b: Multi organ dysfunction Grade V Death of a patient Suffix 'd': If the patient suffers from a complication at the time of discharge, the suffix "d" (for 'disability') is added to the respective grade of complication. This label indicates the need for a follow-up to fully evaluate the complication

Any complications equal to or greater than grade III, will be labeled as Severe adverse events (SAEs). All SAEs will be managed as per the hospital protocol. Any such events will be reviewed thoroughly and the factor responsible for SAE will be identified so as to prevent them in future.

6. Statistical consideration Both descriptive and inferential statistics will be used. The outcome variables will be expressed as frequency and percentage for categorical variables, mean with standard deviation; median and interquartile range for continuous variables. The association between the categorical outcome variables will be sought using Chi square test. The comparison of difference in mean score between the same group will be performed by paired T test while the comparison of means between two different groups will be done by independent T test.

7. Data Management

The data will be collected by the principal investigator. The validity and fidelity of the data will be periodically monitored by the DSMB. The data will be collected using preformed proforma and PFDI-20. The collected data will be coded and entered in Ms Excel spreadsheet. The data will be then analyzed using SPSS version. The primary outcome will be analyzed according to original treatment assignment plan (Per protocol analysis). The success will also be analyzed according to intention to treat analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Women with stage 2-4 pelvic organ prolapse with or without uterus planned for vaginal surgery
2. Women requiring concomitant surgical procedure for incontinence as needed

Exclusion Criteria:

1. Women with pelvic organ prolapse planned for abdominal surgery
2. Women undergoing uterus preserving surgery for pelvic organ prolapse
3. Women undergoing Fothergill's repair/ Obliterative procedures
4. Pregnant or postpartum women with prolapse
5. Women refusing consent to participate in the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Success rate of SSLF and USLS for apical suspension | 6 months after surgery
  Success will be defined as absence of any of the following
  1. Stage II or greater apical compartment prolapse
  2. Awareness of bulge symptoms confirmed by affirmative response to question number 3 of PFDI-20.
  3. Need of additional treatment for prolapse (ring pessary, repeat surgery)
Success rate of SSLF and USLS for apical suspension | 12 months after surgery
  Success will be defined as absence of any of the following
  1. Stage II or greater apical compartment prolapse
  2. Awareness of bulge symptoms confirmed by affirmative response to question number 3 of PFDI-20.
  3. Need of additional treatment for prolapse (ring pessary, repeat surgery)

SECONDARY OUTCOMES:
Perioperative outcomes | 1 week of surgery
  includes: Duration of surgery Intraoperative blood loss Duration of catheterization Duration of Hospital stay
Complications | during surgery, follow up at 6 month and 12 month
  Bladder, ureteric or bowel injury, neurological injury, vascular injury Urinary retention, Vault hematoma, Dyspareunia
postoperative PFDI- 20 score | 6 months and 12 months post surgery
  change in PFDI-20 score from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Tulasa Basnet, MD, Principal Investigator — B.P. Koirala Institute of Health Sciences; Mohan Chandra Regmi, MD, Study Chair — B.P. Koirala Institute of Health Sciences; Baburam Dixit Thapa, MD, Principal Investigator — B.P. Koirala Institute of Health Sciences; Aparna Hegde, MD, Principal Investigator — Grant Medical College, Mumbai

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared till the end of the study. The study protocol will be published prior to publication of the research findings. All the relevant data will be shared with final report of the study as supplementary files.